CLINICAL TRIAL: NCT04040673
Title: Evaluation of the Role of Vibrational Spectroscopy in the Diagnosis of Premalignant and Malignant Disease of the Thyroid RAFTER (RAman For Thyroid cancER)
Brief Title: RAman For Thyroid cancER
Acronym: RAFTER
Status: Not yet recruiting | Type: Observational
Sponsor: Gloucestershire Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Alex Dudgeon, Post-Doctoral Research Fellow, Gloucestershire Hospitals NHS Foundation Trust
Other Study IDs: 18/044/GHT; 245612 (Other: IRAS); 18/LO/1545 (Other: REC)
Record Dates: First submitted 2019-07-29; First posted 2019-08-01 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Thyroid Diseases; Thyroid Cancer
Keywords: cancer; Raman; thyroid
MeSH Terms: conditions — Thyroid Diseases; Thyroid Neoplasms; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Normal benign: participants with normal benign nodules (no cancer)
  Interventions: Procedure: thyroid lobectomy; Device: Raman spectroscopy probe measurement
- Follicular thyroid cancer: participants with follicular thyroid cancer
  Interventions: Procedure: thyroid lobectomy; Device: Raman spectroscopy probe measurement
- Papillary thyroid cancer: participants with papillary thyroid cancer
  Interventions: Procedure: thyroid lobectomy; Device: Raman spectroscopy probe measurement
- Anaplastic thyroid cancer: participants with anaplastic thyroid cancer
  Interventions: Procedure: thyroid lobectomy; Device: Raman spectroscopy probe measurement
- Medullary thyroid cancer: participants with medullary thyroid cancer
  Interventions: Procedure: thyroid lobectomy; Device: Raman spectroscopy probe measurement

INTERVENTIONS:
Procedure: thyroid lobectomy — routine surgical removal of thyroid for biopsy
  Other Names: thyroid nodule removal
Device: Raman spectroscopy probe measurement — The measurement of Raman spectra from the excised tissue

SUMMARY:
Ex vivo vibrational spectroscopy (VS), including Raman spectroscopy (RS) of thyroid tissue samples, collected from patients undergoing routine diagnostic thyroid biopsies for diagnosis of potential thyroid cancer. Raman spectra are to be correlated with consensus histopathology and clinical outcomes. Multivariate analysis to be used to evaluate the classification accuracy of VS ex vivo.

DETAILED DESCRIPTION:
The Investigators (The Biophotonics Research Unit, University of Exeter and University of Bristol) have developed these "smart needle" probes, consisting of fibre-optics within a fine needle for investigating cancer below the skin's surface. It is difficult to create a sensitive probe to fit inside a needle; however, The Investigators have demonstrated this approach in lymph node tissue samples from 68 patients in the laboratory, where The Investigators showed that our probe could detect cancer with a high level of accuracy.

Following on from our success with lymph nodes The Investigators wish to trial our smart needle on excised thyroid to demonstrate the device in another ENT cancer. Earlier studies have shown that thyroid cancer can be diagnosed using RS under a microscope with an accuracy greater than 78%.9 By eliminating the need for unnecessary surgery by diagnosis with our device, The Investigators will minimise the risk to patients, eliminate delays in obtaining results and reduce the cost of surgery and overnight stay in the hospital. The Investigators wish to advance this device closer to the clinic for a new cancer to improve the patient care pathway and remove the need for unnecessary surgery, by facilitating the work of the one-stop ENT diagnostic outpatient clinics.

The study consists of measuring spectra of new tissue taken during routine diagnostic surgical thyroid lobectomy.

New tissue for this project will be collected during routine biopsy will be rapidly analysed by a spectrometer before proceeding with conventional histopathological analysis. The new tissue will consist of thyroid and adjacent tissue biopsies. No additional tissue will be taken for this research, The Investigators only plan to measure samples taken during routine diagnosis in under 5 minutes, before passing the sections back to the surgical team for routine histopathological analysis.

Anonymous background information relevant to known risk factors, family history and details of any treatment, menopausal status, details relevant medical procedures, and any treatment for thyroid cancer will be provided with the samples. An example of the report can be found in Appendix 3. Tissue specimens taken during routine clinical care are to be subjected to ex vivo vibrational spectroscopic analysis immediately prior to being sent for routine histopathological analysis. Vibrational spectra are to be correlated with consensus histopathology of adjacent sections. Multivariate analysis is to be used to evaluate the classification accuracy of VS ex vivo. The vibrational spectra will be assessed for both prognostic as well as diagnostic information.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing routine diagnostic thyroid biopsy at surgery

Exclusion Criteria:

* Patients are unable to provide informed consent.
* Patients not attending for standard diagnostic biopsy for thyroid cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients attending for routine diagnostic biopsy
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Test the Raman needle probe on freshly exised tissue | 1 year
  Measure Raman spectra and match with histopathology. Perform leave-one-out analysis to measure performance of diagnosis of Raman spectroscopy

SECONDARY OUTCOMES:
Calculate diagnostic performance of Raman spectroscopy probe for thyroid cancer | 1 year
  Diagnostic performance (specificity and sensitivity) of Raman spectroscopy (RS) for differentiation of thyroid cancer vs normal benign (no cancer).
  Diagnostic performance of RS for differentiation of thyroid cancer types.
  * Papillary thyroid cancer
  * Follicular thyroid cancer
  * Anaplastic thyroid cancer
  * Medullary thyroid cancer

CONTACTS AND LOCATIONS:
Locations (1):
- Biophotonics Research Unit, Gloucester, Gloucestershire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Pathology reports will be linked using a pseudo-anonymous unique study identifier

REFERENCES:
- [Background] Kamran SC, Marqusee E, Kim MI, Frates MC, Ritner J, Peters H, Benson CB, Doubilet PM, Cibas ES, Barletta J, Cho N, Gawande A, Ruan D, Moore FD Jr, Pou K, Larsen PR, Alexander EK. Thyroid nodule size and prediction of cancer. J Clin Endocrinol Metab. 2013 Feb;98(2):564-70. doi: 10.1210/jc.2012-2968. Epub 2012 Dec 28. PMID 23275525
- [Background] Jenkins CA, Lewis PD, Dunstan PR, Harris DA. Role of Raman spectroscopy and surface enhanced Raman spectroscopy in colorectal cancer. World J Gastrointest Oncol. 2016 May 15;8(5):427-38. doi: 10.4251/wjgo.v8.i5.427. PMID 27190582
- [Background] Feng X, Moy AJ, Nguyen HTM, Zhang J, Fox MC, Sebastian KR, Reichenberg JS, Markey MK, Tunnell JW. Raman active components of skin cancer. Biomed Opt Express. 2017 May 4;8(6):2835-2850. doi: 10.1364/BOE.8.002835. eCollection 2017 Jun 1. PMID 28663910
- [Background] Crow P, Barrass B, Kendall C, Hart-Prieto M, Wright M, Persad R, Stone N. The use of Raman spectroscopy to differentiate between different prostatic adenocarcinoma cell lines. Br J Cancer. 2005 Jun 20;92(12):2166-70. doi: 10.1038/sj.bjc.6602638. PMID 15928665
- [Background] Rau JV, Fosca M, Graziani V, Taffon C, Rocchia M, Caricato M, Pozzilli P, Onetti Muda A, Crescenzi A. Proof-of-concept Raman spectroscopy study aimed to differentiate thyroid follicular patterned lesions. Sci Rep. 2017 Nov 2;7(1):14970. doi: 10.1038/s41598-017-14872-1. PMID 29097686

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/73/NCT04040673/Prot_ICF_000.pdf